CLINICAL TRIAL: NCT02927210
Title: Injectable DMAU for Male Contraception: Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of Single IM or SC DMAU Injection Dose Escalation Study in Healthy Male Volunteers
Brief Title: Injectable DMAU for Male Contraception in Healthy Male Volunteers (CCN015)
Acronym: DMAU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kimberly Myer (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Kimberly Myer, Program Director, Premier Research
Organization: Premier Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CCN015; HHSN275201200002I (Other Grant/Funding Number: NICHD Contract. This is not a grant but a contract.)
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Men; Male Contraception
Keywords: Healthy Men; Male Contraception; Androgen; Dimethandrolone
MeSH Terms: interventions — dimethandrolone-undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo injections that look like the DMAU injections but with no active ingredients
  Interventions: Drug: Placebo
- Dimethandrolone Undecanoate (Experimental): Single doses of DMAU administered via injection intramuscularly (IM - 80 mg, 240 mg, 480 mg, and 800 mg) or administered subcutaneously (SC - 50 mg, 100 mg and 200 mg)
  Interventions: Drug: Dimethandrolone Undecanoate

INTERVENTIONS:
Drug: Dimethandrolone Undecanoate — Single doses of DMAU in castor oil/benzyl benzoate injections intramuscularly (IM) (80 mg, 240 mg, 480 mg, and 800 mg) or administered subcutaneously (SC) (50 mg, 100 mg and 200 mg).
  Other Names: DMAU
  Arms: Dimethandrolone Undecanoate
Drug: Placebo — Placebo injections that look like the DMAU injections but with no active ingredients
  Arms: Placebo

SUMMARY:
This is a Phase I multicenter, double-blind, single dose, dose-ranging study, in healthy men to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of Dimethandrolone Undecanoate (DMAU) administered as an intramuscular or subcutaneous injection.

DETAILED DESCRIPTION:
This single dose, dose-ranging study will be conducted in two centers: the Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center and the University of Washington.

Single doses of DMAU in castor oil/benzyl benzoate injections intramuscularly (IM) (80 mg, 240 mg, 480 mg, and 800 mg) or administered subcutaneously (SC) (50 mg, 100 mg and 200 mg) were selected for this dose-escalating study. Twelve subjects will complete this study at each of the DMAU doses (10 on DMAU and 2 on placebo injections) yielding a total of 84 completed subjects (70 on DMAU and 14 on placebo) across both sites. Safety will be assessed in all subjects and recovery will be assessed in two subjects receiving lower doses, either IM or SC, before additional men receive higher doses of IM or SC of DMAU. In addition to safety and tolerability, suppression of serum T, E2, gonadotropins, and SHBG will be assessed as secondary pharmacodynamic (PD) endpoints. PK of DMAU and DMA will be assessed through blood draws done at each visit. Suppression of spermatogenesis will be assessed with semen analysis.

DMAU injections will be administered at the study site by research nurses or physicians. For intramuscular injections, the staff will inject DMAU in castor oil into the gluteal region following standard procedures for intramuscular steroid injection. Abdominal subcutaneous injections will follow standard subcutaneous procedures. The subject will be observed for at least 30 minutes before release from the study site.

ELIGIBILITY:
Inclusion Criteria:

Men who meet all the following criteria are eligible for enrollment in the trial:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening.
2. 18 to 50 years of age (inclusive) at the time of the enrollment visit.
3. BMI ≤ 33 calculated as weight in kg/ (height in m2).
4. Weight ≥60 kg.
5. No history of hormonal therapy use in the three months prior to the first screening visit.
6. Agree to use a recognized effective method of contraception with any female partner (i.e. at a minimum, barrier plus an additional method of contraception) during the course of the study treatment and recovery phases until recovery is confirmed and study exit occurs.
7. Subjects will refrain from donating blood or plasma during the study period.
8. Subjects will be advised to refrain from excessive alcoholic consumption during the study period. (No more than 15 drinks per week and no alcohol consumption within 24 hours of a study visit.)
9. No known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
10. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form.

12. Subjects will be advised to refrain from major changes in their level of exercise during the study period.

Exclusion Criteria:

Men who meet any of the following criteria are NOT eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within the 30 days prior to the first screening visit.
2. Men not living in the catchment area of the clinic or within a reasonable distance from the study site.
3. Clinically significant abnormal physical and laboratory findings at screening.
4. Elevated PSA (levels ≥ 2.5 ng/mL) at screening, according to local laboratory normal values.
5. Abnormal serum chemistry values at screening, according to local laboratory reference ranges that indicate liver or kidney dysfunction or that may be considered clinically significant. In addition, the following upper limits will be observed: fasting bilirubin less than 2 mg/dL, cholesterol less than 221 mg/dL, and fasting triglycerides less than 201 mg/dL.
6. Abnormal semen analyses or abnormal semen concentration as defined by the WHO semen manual.
7. Use of androgens within 3 months before first screening visit except for long acting testosterone injections (e.g. Testosterone undecanoate) which will require a wash out period of 6 months prior to screening.
8. Ongoing use of body building substances including nutritional supplements.
9. Systolic BP > 130 mm Hg and Diastolic blood pressure BP > 80 and mm Hg; Blood pressure (BP) will be taken 3 times at 5 - minute intervals and the mean of all measurements be used to determine eligibility).
10. Clinically significant abnormal EKG or a QTc interval of > 450 msec.
11. PHQ-9 score of 15 or above.
12. History of hypertension, including hypertension controlled with treatment.
13. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
14. Benign or malignant liver tumors; active liver disease.
15. History of breast carcinoma.
16. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease.
17. Known history of cardiovascular, renal, hepatic or prostatic disease or significant psychiatric illness.
18. Positive serology for active Hepatitis (not immunization-related serology) or HIV at screening visit.
19. A serious systemic disease such as diabetes mellitus or obesity (body weight greater than BMI >33 kg/m2 as above).
20. History of known, untreated sleep apnea.

22. Partner is known to be pregnant. 23. Men desiring fertility within the first seven months of study participation.

24. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine. Exclusion is due to the potential of testing positive for androgens that may occur from their study participation coupled with the unknown efficacy (i.e. duration of positive testing) from a single injection.

26. Use of sex steroids or medications which might interfere with steroid metabolism (i.e. ketoconazole, finasteride, oral corticosteroids, dutasteride and statins).

27. Use of medications that will interfere or interact with DMAU.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in sexual function (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) using the psychosexual daily questionnaire | 5-7 months
Changes from baseline in mood (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) using the Patient Health Questionnaire-9 | 5-7 months
Changes from baseline in sodium (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in potassium (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in chloride (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in bicarbonate (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in fasting glucose (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in blood urea nitrogen (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in creatinine (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in calcium (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in total bilirubin (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in alkaline phosphatase (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in alanine aminotransferase (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in aspartate transaminase (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in albumin (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in blood pressure (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in pulse (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in respiratory rate (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months
Changes from baseline in body mass index (safety and tolerability) with a single IM or SC injection of escalating doses of Dimethandrolone Undecanoate (DMAU) | 5-7 months

SECONDARY OUTCOMES:
Pharmacokinetics of DMAU and DMA using AUC (0-t, where t is the last time-point with measurable concentration) | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of serum Testosterone (T) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of Dihydrotestosterone (DHT) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of Estradiol (E2) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of Follicle Stimulating Hormone (FSH) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of Luteinizing Hormone (LH) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of Sex Hormone Binding Globulin (SHBG) using mean values at each visit | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of serum T using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of serum T using percentage of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of DHT using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of DHT using percentage of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of E2 using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of E2 using percentage of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of FSH using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of FSH using of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of LH using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of LH using percentage of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of SHBG using number of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Pharmacodynamics of DMAU by assessing the suppression of SHBG using percentage of subjects with FSH and LH ≤ 1.0 IU/L | 5-7 months
Suppression of spermatogenesis as assessed by semen analyses using number of subjects with sperm concentration <1 million (M)/mL | 5-7 months
Suppression of spermatogenesis as assessed by semen analyses using percentage of subjects with sperm concentration <1 million (M)/mL | 5-7 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Stephanie Page Page, MD, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Washington Medical Center & Health Sciences, Seattle, Washington

REFERENCES:
- [Background] Attardi BJ, Engbring JA, Gropp D, Hild SA. Development of dimethandrolone 17beta-undecanoate (DMAU) as an oral male hormonal contraceptive: induction of infertility and recovery of fertility in adult male rabbits. J Androl. 2011 Sep-Oct;32(5):530-40. doi: 10.2164/jandrol.110.011817. Epub 2010 Dec 16. PMID 21164142
- [Background] Attardi BJ, Hild SA, Koduri S, Pham T, Pessaint L, Engbring J, Till B, Gropp D, Semon A, Reel JR. The potent synthetic androgens, dimethandrolone (7alpha,11beta-dimethyl-19-nortestosterone) and 11beta-methyl-19-nortestosterone, do not require 5alpha-reduction to exert their maximal androgenic effects. J Steroid Biochem Mol Biol. 2010 Oct;122(4):212-8. doi: 10.1016/j.jsbmb.2010.06.009. Epub 2010 Jun 25. PMID 20599615
- [Background] Attardi BJ, Marck BT, Matsumoto AM, Koduri S, Hild SA. Long-term effects of dimethandrolone 17beta-undecanoate and 11beta-methyl-19-nortestosterone 17beta-dodecylcarbonate on body composition, bone mineral density, serum gonadotropins, and androgenic/anabolic activity in castrated male rats. J Androl. 2011 Mar-Apr;32(2):183-92. doi: 10.2164/jandrol.110.010371. Epub 2010 Aug 26. PMID 20798389
- [Background] Attardi BJ, Hild SA, Reel JR. Dimethandrolone undecanoate: a new potent orally active androgen with progestational activity. Endocrinology. 2006 Jun;147(6):3016-26. doi: 10.1210/en.2005-1524. Epub 2006 Feb 23. PMID 16497801
- [Background] Attardi BJ, Pham TC, Radler LC, Burgenson J, Hild SA, Reel JR. Dimethandrolone (7alpha,11beta-dimethyl-19-nortestosterone) and 11beta-methyl-19-nortestosterone are not converted to aromatic A-ring products in the presence of recombinant human aromatase. J Steroid Biochem Mol Biol. 2008 Jun;110(3-5):214-22. doi: 10.1016/j.jsbmb.2007.11.009. PMID 18555683
- [Background] Cook CE, Kepler JA. 7alpha,11beta-Dimethyl-19-nortestosterone: a potent and selective androgen response modulator with prostate-sparing properties. Bioorg Med Chem Lett. 2005 Feb 15;15(4):1213-6. doi: 10.1016/j.bmcl.2004.11.076. PMID 15686944
- [Background] Cummings DE, Kumar N, Bardin CW, Sundaram K, Bremner WJ. Prostate-sparing effects in primates of the potent androgen 7alpha-methyl-19-nortestosterone: a potential alternative to testosterone for androgen replacement and male contraception. J Clin Endocrinol Metab. 1998 Dec;83(12):4212-9. doi: 10.1210/jcem.83.12.5324. PMID 9851754
- [Background] Frey-Wettstein M, Craddock CG. Testosterone-induced depletion of thymus and marrow lymphocytes as related to lymphopoiesis and hematopoiesis. Blood. 1970 Mar;35(3):257-71. No abstract available. PMID 4908652
- [Background] Gu Y, Liang X, Wu W, Liu M, Song S, Cheng L, Bo L, Xiong C, Wang X, Liu X, Peng L, Yao K. Multicenter contraceptive efficacy trial of injectable testosterone undecanoate in Chinese men. J Clin Endocrinol Metab. 2009 Jun;94(6):1910-5. doi: 10.1210/jc.2008-1846. Epub 2009 Mar 17. PMID 19293262
- [Background] Gu YQ, Wang XH, Xu D, Peng L, Cheng LF, Huang MK, Huang ZJ, Zhang GY. A multicenter contraceptive efficacy study of injectable testosterone undecanoate in healthy Chinese men. J Clin Endocrinol Metab. 2003 Feb;88(2):562-8. doi: 10.1210/jc.2002-020447. PMID 12574181
- [Background] Hild SA, Attardi BJ, Koduri S, Till BA, Reel JR. Effects of synthetic androgens on liver function using the rabbit as a model. J Androl. 2010 Sep-Oct;31(5):472-81. doi: 10.2164/jandrol.109.009365. Epub 2010 Apr 8. PMID 20378929
- [Background] Ilani N, Roth MY, Amory JK, Swerdloff RS, Dart C, Page ST, Bremner WJ, Sitruk-Ware R, Kumar N, Blithe DL, Wang C. A new combination of testosterone and nestorone transdermal gels for male hormonal contraception. J Clin Endocrinol Metab. 2012 Oct;97(10):3476-86. doi: 10.1210/jc.2012-1384. Epub 2012 Jul 12. PMID 22791756
- [Background] Lee KK, Berman N, Alexander GM, Hull L, Swerdloff RS, Wang C. A simple self-report diary for assessing psychosexual function in hypogonadal men. J Androl. 2003 Sep-Oct;24(5):688-98. doi: 10.1002/j.1939-4640.2003.tb02728.x. PMID 12954659
- [Background] Kaminetsky J, Jaffe JS, Swerdloff RS. Pharmacokinetic Profile of Subcutaneous Testosterone Enanthate Delivered via a Novel, Prefilled Single-Use Autoinjector: A Phase II Study. Sex Med. 2015 Sep 17;3(4):269-79. doi: 10.1002/sm2.80. eCollection 2015 Dec. PMID 26797061
- [Background] Keenan CM, Vidal JD. Standard morphologic evaluation of the heart in the laboratory dog and monkey. Toxicol Pathol. 2006;34(1):67-74. doi: 10.1080/01926230500369915. PMID 16507546
- [Background] Kumar N, Didolkar AK, Monder C, Bardin CW, Sundaram K. The biological activity of 7 alpha-methyl-19-nortestosterone is not amplified in male reproductive tract as is that of testosterone. Endocrinology. 1992 Jun;130(6):3677-83. doi: 10.1210/endo.130.6.1597164.
- [Background] Kumar N, Suvisaari J, Tsong YY, Aguillaume C, Bardin CW, Lahteenmaki P, Sundaram K. Pharmacokinetics of 7 alpha-methyl-19-nortestosterone in men and cynomolgus monkeys. J Androl. 1997 Jul-Aug;18(4):352-8. PMID 9283946
- [Background] Malhotra A, Buttrick P, Scheuer J. Effects of sex hormones on development of physiological and pathological cardiac hypertrophy in male and female rats. Am J Physiol. 1990 Sep;259(3 Pt 2):H866-71. doi: 10.1152/ajpheart.1990.259.3.H866. PMID 2144404
- [Background] Marsh JD, Lehmann MH, Ritchie RH, Gwathmey JK, Green GE, Schiebinger RJ. Androgen receptors mediate hypertrophy in cardiac myocytes. Circulation. 1998 Jul 21;98(3):256-61. doi: 10.1161/01.cir.98.3.256. PMID 9697826
- [Background] Meriggiola MC, Costantino A, Bremner WJ, Morselli-Labate AM. Higher testosterone dose impairs sperm suppression induced by a combined androgen-progestin regimen. J Androl. 2002 Sep-Oct;23(5):684-90. PMID 12185103
- [Background] Morgentaler A, Dobs AS, Kaufman JM, Miner MM, Shabsigh R, Swerdloff RS, Wang C. Long acting testosterone undecanoate therapy in men with hypogonadism: results of a pharmacokinetic clinical study. J Urol. 2008 Dec;180(6):2307-13. doi: 10.1016/j.juro.2008.08.126. Epub 2008 Oct 18. PMID 18930255
- [Background] Rothman MS, Carlson NE, Xu M, Wang C, Swerdloff R, Lee P, Goh VH, Ridgway EC, Wierman ME. Reexamination of testosterone, dihydrotestosterone, estradiol and estrone levels across the menstrual cycle and in postmenopausal women measured by liquid chromatography-tandem mass spectrometry. Steroids. 2011 Jan;76(1-2):177-82. doi: 10.1016/j.steroids.2010.10.010. Epub 2010 Nov 9. PMID 21070796
- [Background] Surampudi P, Page ST, Swerdloff RS, Nya-Ngatchou JJ, Liu PY, Amory JK, Leung A, Hull L, Blithe DL, Woo J, Bremner WJ, Wang C. Single, escalating dose pharmacokinetics, safety and food effects of a new oral androgen dimethandrolone undecanoate in man: a prototype oral male hormonal contraceptive. Andrology. 2014 Jul;2(4):579-587. doi: 10.1111/j.2047-2927.2014.00216.x. Epub 2014 May 2. PMID 24789057
- [Background] Swerdloff RS, Wang C, Cunningham G, Dobs A, Iranmanesh A, Matsumoto AM, Snyder PJ, Weber T, Longstreth J, Berman N. Long-term pharmacokinetics of transdermal testosterone gel in hypogonadal men. J Clin Endocrinol Metab. 2000 Dec;85(12):4500-10. doi: 10.1210/jcem.85.12.7045. PMID 11134099
- [Background] Vermeulen A, Verdonck L, Kaufman JM. A critical evaluation of simple methods for the estimation of free testosterone in serum. J Clin Endocrinol Metab. 1999 Oct;84(10):3666-72. doi: 10.1210/jcem.84.10.6079. PMID 10523012
- [Background] von Eckardstein S, Noe G, Brache V, Nieschlag E, Croxatto H, Alvarez F, Moo-Young A, Sivin I, Kumar N, Small M, Sundaram K; International Committee for Contraception Research, The Population Council. A clinical trial of 7 alpha-methyl-19-nortestosterone implants for possible use as a long-acting contraceptive for men. J Clin Endocrinol Metab. 2003 Nov;88(11):5232-9. doi: 10.1210/jc.2002-022043. PMID 14602755
- [Background] Wang C, Catlin DH, Demers LM, Starcevic B, Swerdloff RS. Measurement of total serum testosterone in adult men: comparison of current laboratory methods versus liquid chromatography-tandem mass spectrometry. J Clin Endocrinol Metab. 2004 Feb;89(2):534-43. doi: 10.1210/jc.2003-031287. PMID 14764758
- [Background] Wang C, Harnett M, Dobs AS, Swerdloff RS. Pharmacokinetics and safety of long-acting testosterone undecanoate injections in hypogonadal men: an 84-week phase III clinical trial. J Androl. 2010 Sep-Oct;31(5):457-65. doi: 10.2164/jandrol.109.009597. Epub 2010 Feb 4. PMID 20133964
- [Background] Wang C, Shiraishi S, Leung A, Baravarian S, Hull L, Goh V, Lee PW, Swerdloff RS. Validation of a testosterone and dihydrotestosterone liquid chromatography tandem mass spectrometry assay: Interference and comparison with established methods. Steroids. 2008 Dec 12;73(13):1345-52. doi: 10.1016/j.steroids.2008.05.004. Epub 2008 May 21. PMID 18579171
- [Background] Wang C, Swerdloff R, Kipnes M, Matsumoto AM, Dobs AS, Cunningham G, Katznelson L, Weber TJ, Friedman TC, Snyder P, Levine HL. New testosterone buccal system (Striant) delivers physiological testosterone levels: pharmacokinetics study in hypogonadal men. J Clin Endocrinol Metab. 2004 Aug;89(8):3821-9. doi: 10.1210/jc.2003-031866. PMID 15292312
- [Background] Weinbauer GF, Gockeler E, Nieschlag E. Testosterone prevents complete suppression of spermatogenesis in the gonadotropin-releasing hormone antagonist-treated nonhuman primate (Macaca fascicularis). J Clin Endocrinol Metab. 1988 Aug;67(2):284-90. doi: 10.1210/jcem-67-2-284. PMID 3292557
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] World Health Organization Task Force on Methods for the Regulation of Male Fertility. Contraceptive efficacy of testosterone-induced azoospermia and oligozoospermia in normal men. Fertil Steril. 1996 Apr;65(4):821-9. PMID 8654646